CLINICAL TRIAL: NCT04962282
Title: Research on Influencing Factors of Compliance of Spinal Exercise Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019385
Record Dates: First submitted 2021-06-27; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Non-specific Chronic Low Back Pain
Keywords: Non-specific Chronic Low Back Pain; Home-based Exercise Therapy; Adherence

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group 1: Follow-up by telephone for researching compliance of patients receiving exercise prescriptions
  Interventions: Other: Follow-up by telephone

INTERVENTIONS:
Other: Follow-up by telephone — Studies have shown that the compliance of patients at 8-12 weeks reaches a peak, so this time node is the most suitable time node to investigate compliance. Telephone follow-up is irreplaceable convenience, so the telephone follow-up survey of patient compliance with exercise prescriptions is The most feasible method The purpose of the telephone follow-up is to 1. Investigate the compliance of the patients; 2. Make the patients fill out a self-made research compliance scale influencing factors through the telephone.The purpose of the telephone follow-up is to 1. Investigate the compliance of the patients; 2. Make the patients fill out a self-made research compliance scale influencing factors through the telephone.

SUMMARY:
Explore the many factors that affect the compliance of home exercise therapy in patients with non-specific chronic low back pain, establish a theoretical model of the factors affecting compliance behavior, in order to guide rehabilitation clinical practice, and improve the compliance of patients with non-specific chronic low back pain to home exercise prescriptions.

DETAILED DESCRIPTION:
ABSTRACT Objective: To achieve more information and establish better guidance for the clinical practice of rehabilitation, to improve the adherence of non-specific chronic low back pain patients with home-based exercise prescription by exploring the factors that affect the adherence of patients, and by building a theoretical model of adherence influencing factors.

Method: From February 2019 to August 2019, 39 patients were diagnosed as non-specific chronic low back pain and prescribed home-based exercise prescription in the Department of rehabilitation medicine of Peking University Third Hospital. They were recruited by criterion-based sampling and had face-to-face exercise therapy guidance from the same physiotherapist. We have a semi-structured 20-40 minutes telephone interview 2-3 months later. The conversation was recorded with the consent of the patients, then the recorded content was documented as text data. By the patient's exercise type, intensity, duration and frequency, the patient adherence was classified as complete adherent, partial adherent and complete not adherent. The qualitative research method was used to analyze the data under the guidance of grounded theory with the help of qualitative analysis software NVivo. NVivo was used to encode the text data of patient's conversation in three levels, and the themes were extracted to explain the causes of adherence.

Result: Of the 39 patients interviewed, 32 responded to the interview, with a response rate of 82.0%. The average age of these 32 responded patients was 48.8±18.6 years old. There were 9 males (28.1%) and 23 females (71.9%). There were 4 complete adherent patients, 5 not adherent, and 23 partial adherent (including 14 giving up halfway and 9 intermittent exercise). The open coding got 19 initial sub-categories; then axial coding classified 19 initial sub-categories into five main categories, namely health belief, self-efficacy, exercise prescription, self-management and family support. Selective coding classified health belief and self-efficacy as "internal environment", while exercise prescription and family support as "external environment". Based on this discovery, two theories are established: (1) patients' "self-management" ability is the internal motivation of adherence behavior; (2) the "internal environment" and "external environment" play a regulatory role in adherence behavior.

Conclusion: Patients' adherence behavior is directly affected by the ability of self-management and tends to be standardized under the regulation of good internal and external environment. Regular follow-up, health education and adjusting the structure of exercise prescription are necessary measures to improve patients' adherence.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age from 18 to 80 years old; 2.The clinical diagnosis is non-specific low back pain, the course of disease is ≥12 weeks;

Exclusion Criteria:

* 1.Combined with specific lumbar spine diseases, physical diseases affecting sports 2.Due to mental or psychological abnormalities; refused to accept telephone interviews; 3.Failed to answer the interview call for 3 consecutive times;

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: From February 2019 to August 2019, due to recurrent low back pain, he was treated in the Department of Rehabilitation Medicine of Peking University Third Hospital and prescribed home exercise therapy.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
main result 1 | 8 weeks after receiving treatment
  The number of patients with good compliance;
main result 2 | 8 weeks after receiving treatment
  the number of patients with poor compliance
main result 3 | 8 weeks after receiving treatment
  Self-made scale scores in 8 dimensions

CONTACTS AND LOCATIONS:
Locations (1):
- Research on Influencing Factors of Compliance of Spinal Exercise Therapy, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No